CLINICAL TRIAL: NCT02986906
Title: The Long-term Effect for Perineural Injection Therapy for Ulnar Neuropathy at Elbow
Brief Title: Perineural Injection Therapy for Ulnar Neuropathy at Elbow
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Yung-Tsan Wu, Attending Physician of Department of Physical Medicine and Rehabilitation, Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PIT for ulnar neuropathy
Record Dates: First submitted 2016-12-06; First posted 2016-12-08 (Estimated); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Ulnar Neuropathy at Elbow
Keywords: ulnar neuropathy at elbow; Dextrose; perineural injection
MeSH Terms: interventions — Glucose; Ultrasonography

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 5% dextrose (Experimental): The perineural injection with 5% dextrose is a new and potential treatment for peripheral entrapment neuropathy
  Interventions: Drug: 5% dextrose; Device: Ultrasound
- 2cc 0.9% normal saline+3cc Triamcinolone (30mg) (Active Comparator): The Ultrasound-guided injection with 2cc 0.9% normal saline+3cc Triamcinolone (30mg)
  Interventions: Drug: 2cc 0.9% normal saline+3cc Triamcinolone (30mg); Device: Ultrasound

INTERVENTIONS:
Drug: 5% dextrose — Ultrasound-guided 5cc 5% dextrose injection between medial epicondyle and ulnar nerve
  Arms: 5% dextrose
Drug: 2cc 0.9% normal saline+3cc Triamcinolone (30mg) — Ultrasound-guided 2cc 0.9% normal saline+3cc Triamcinolone (30mg) injection between medial epicondyle and ulnar nerve
  Arms: 2cc 0.9% normal saline+3cc Triamcinolone (30mg)
Device: Ultrasound — The ultrasound was used for injection guidance

SUMMARY:
Ulnar neuropathy at elbow (UNE) is the second common peripheral entrapment neuropathy. Although many conservative managements of UNE, the effectiveness of these methods are unsatisfied especial the moderate degree of UNE. Recently, ultrasound-guided perineural injection therapy (PIT) with 5% dextrose is progressively applicated for clinical treatment for entrapment neuropathy. However, current studies have not proved the effects of PIT on peripheral neuropathy because these studies enrolled small number of patients and lacked controlled design. We design a randomized, double-blind, controlled trail to assess the effect after ultrasound-guided PIT with 5% dextrose in patients with mild and moderate UNE.

DETAILED DESCRIPTION:
After obtaining written informed consent, 40 patients, clinically diagnosed with mild or moderate UNE were randomized into intervention or control group. Participants in intervention group received one-session of ultrasound-guided PIT injection with 5cc. 5% dextrose and control group received 2cc 0.9% normal saline+3cc Triamcinolone (30mg) (total 5 cc) ultrasound-guided PIT injection. The primary outcome is Disabilities of the Arm, Shoulder and Hand (DASH) and secondary outcomes include visual analog scale (VAS), cross-sectional area (CSA) of the ulnar nerve, motor nerve conduction velocity of the ulnar nerve, and strength of palmer finger pinch and grasp. The evaluation was performed pretreatment as well as on the 1st, 3rd and 6th month after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20-80 year-old.
* Diagnosis was confirmed using an electrophysiological study

Exclusion Criteria:

* Cancer
* Coagulopathy
* Pregnancy
* Inflammation status
* Cervical radiculopathy
* Polyneuropathy, brachial plexopathy
* Thoracic outlet syndrome
* Previously undergone wrist surgery or steroid injection for ulnar neuropathy

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Change from pain on 1st, 3rd, 6th month after injection | Pre-treatment, 1st, 3rd, 6th month after injection
  Digital pain severity or paresthesia/dysthesia was evaluated using visual analog scale (VAS). Pain score scale ranged from 0 to 10, with 10 indicating the most severe pain.

SECONDARY OUTCOMES:
Change from severity of symptoms and functional status on 1st, 3rd, 6th month after injection | Pre-treatment, 1st, 3rd, 6th month after injection
  Taiwan Disabilities of the Arm, Shoulder and Hand (DASH) contains 11-item disability/symptom scale and each item has five levels of response scoring from 1 to 5. The higher score means more disability or severer symptoms.
Change from nerve conduction velocity on 1st, 3rd, 6th month after injection | Pre-treatment, 1st, 3rd, 6th month after injection
  Nerve motor conduction velocity of the ulnar nerve before treatment and multiple time frame after treatment.
Change from cross-sectional area on 1st, 3rd, 6th month after injection | Pre-treatment, 1st, 3rd, 6th month after injection
  Using the musculoskeletal sonogram to measure the cross-sectional area of the ulnar nerve before treatment and multiple time frame after treatment.
Change from palmer finger pinch and grasp on 1st, 3rd, 6th month after injection | Pre-treatment, 1st, 3rd, 6th month after injection
  The palmer finger pinch and grasp strength was measured using dynamometer (Fabrication Enterprises Inc., USA) before treatment and multiple time frame after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Yung-Tsan Wu, MD, Principal Investigator — Department of Physical Medicine and Rehabilitation, Tri-Service General Hospital
Locations (1):
- Department of Physical Medicine and Rehabilitation, Tri-Service General Hospital, Taipei, Neihu District, Taiwan

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Chang KV, Hung CY, Ozcakar L. Snapping Thumb and Superficial Radial Nerve Entrapment in De Quervain Disease: Ultrasound Imaging/Guidance Revisited. Pain Med. 2015 Nov;16(11):2214-5. doi: 10.1111/pme.12867. Epub 2015 Jul 27. No abstract available. PMID 26218266
- [Result] Campbell WW, Pridgeon RM, Sahni KS. Short segment incremental studies in the evaluation of ulnar neuropathy at the elbow. Muscle Nerve. 1992 Sep;15(9):1050-4. doi: 10.1002/mus.880150910. PMID 1518514
- [Result] Mulvaney SW. Ultrasound-guided percutaneous neuroplasty of the lateral femoral cutaneous nerve for the treatment of meralgia paresthetica: a case report and description of a new ultrasound-guided technique. Curr Sports Med Rep. 2011 Mar-Apr;10(2):99-104. doi: 10.1249/JSR.0b013e3182110096. PMID 21623291